CLINICAL TRIAL: NCT06761196
Title: Assessing Quality of Life After Breast Cancer Surgery: a Prospective Cohort Study
Brief Title: Quality of Life After Breast Cancer Surgery
Acronym: SOCOM-QoL
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de Colmar (Other)
Responsible Party: Sponsor
Other Study IDs: HCC-009; 2024-A02572-45 (Other: ID-RCB - ANSM)
Record Dates: First submitted 2024-12-12; First posted 2025-01-07 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Surgery; Quality of Life
Keywords: breast cancer; oncoplastic surgery; quality of life; quality of recovery
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Questionnaire — The quality of life measured with different scales (BREAST-Q, EORTC QLQ C30 and BR42)

SUMMARY:
The goal of this observational study is to prospectively collect data on quality of life after oncoplastic breast surgery.

Participants will be followed-up and answer quality of life questionnaire for a duration of 5 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over
* Patient with breast cancer of any stage (including in situ) or healthy individual at high personal risk.
* Patient requiring breast surgery under general anesthesia, whether for therapeutic or prophylactic purposes.
* Patient capable, in the opinion of the investigator, of complying with the requirements and restrictions of the study.
* Patient with a computer, tablet or smartphone connected to the Internet.
* Patient followed in the center on a regular basis according to standard recommendations.

Exclusion Criteria:

* Patient requiring surgical intervention under local anesthesia only.
* Patient requiring surgery for the installation or removal of an chemotherapy implantable port only.
* Patients with a history of cancer other than breast cancer. Patients with a history of cancer more than three years old are eligible if they are treated and considered cured. Patients with a history of cervical carcinoma in situ or non-melanoma skin carcinoma are eligible.
* Impossibility of being subject to regular monitoring for geographical, social or psychological reasons.
* Patient under protective measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2035-09-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life measured with BREAST-Q | From enrollment to the end of 5 years follow-up
  The BREAST-Q is a rigorously developed patient-reported outcome measure for use in cosmetic and reconstructive breast surgery and clinical practice. The BREAST-Q conceptual framework covers 2 domains: quality of life, and patient satisfaction. There is three independent modules developped for breast cancer (mastectomy, breast-conserving therapy, reconstruction).
  A conversion table is used to convert the raw scale summed score into a score from 0 (worst) to 100 (best). Higher scores reflect a better outcome.

SECONDARY OUTCOMES:
Quality of life measured with EORTC QLQ C30 | From enrollment to the end of 5 years follow-up
  The EORTC QLG Core Questionnaire (EORTC QLQ-C30) is a 30-item instrument designed to measure quality of life in all cancer patients.
  The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  Each of the multi-item scales includes a different set of items - no item occurs in more than one scale.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
  Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Quality of life measured with EORTC QLQ-BR42 | From enrollment to the end of 5 years follow-up
  The Breast Cancer Module EORTC QLQ-BR42 is a 42-item instrument designed to measure quality of life in breast cancer patients. It is a supplementary questionnaire module to be employed in conjunction with the QLQ-C30. All of the scales and single item measures range in score from 0 to 100. A high score for the Body Image, Sexual Functioning and Breast Satisfaction scales and for the Future Perspective and Sexual Enjoyment single items represents a high level of functioning, whereas a high score for the Systemic ChemoTherapy Side Effects, Endocrine Symptoms, Arm Symptoms, Breast Symptoms, Hand/foot symptoms/neuropathy, Skeletal Scale and Vaginal Symptoms scales and for the Weight Gain single item represents a high level of symptomatology or problems.
Safety of postoperative period | Form enrollment to the end of 5 years follow-up
  Concerning safety, the endpoint is the duration of Hospital Free Survival (HFS) . HFS is defined as the time interval (in days) without any hospitalization from discharge until death.
Quality of postoperative period | At enrollment aund day 1 and 7 after surgery
  Concerning the quality of the postoperative period, the enpoint is the quality of recovery assessed with the 15-item Quality of Recovery (QoR-15) scale.
  The QoR-15 scale is a validated multidimensional questionnaire that measures postoperative quality of recovery. The scale is ranges from 0 to 150. A higher QoR-15 score reflects higher recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Civils de Colmar, Colmar, France